CLINICAL TRIAL: NCT04192331
Title: A Single-arm Opened Randomized Phase II Study of Nab-paclitaxel Dose Schedual in Advanced Breast Cancer
Brief Title: Nab-paclitaxel Dose Schedual for HER-2 Negative Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Li Huiping, Head of the department of breast oncology, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABC012
Record Dates: First submitted 2019-04-14; First posted 2019-12-10 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: nab-paclitaxel; advanced breast cancer; HER2 negative; dose
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2/3dose strategy (Experimental): HER2 negative advanced breast cancer patient
  Interventions: Drug: nab-paclitaxel regimen1
- 3/4dose strategy (Active Comparator): HER2 negative advanced breast cancer patient
  Interventions: Drug: nab-paclitaxel regimen2

INTERVENTIONS:
Drug: nab-paclitaxel regimen1 — nab-paclitaxel regimen1 means use abraxine with 125mg/m2 at day 1 and day 8 per 21d.
  Other Names: regimen1
  Arms: 2/3dose strategy
Drug: nab-paclitaxel regimen2 — nab-paclitaxel regimen2 means use abraxine with 125mg/m2 at day 1 and day 8 and day 15 per 28d.
  Other Names: regimen2
  Arms: 3/4dose strategy

SUMMARY:
What is the best dosage of Nab-Paclitaxel for chinese? This study would divide patients into two dosage groups: 1) 125mg/m2, 30 minutes intravenous injection, d1, 8, 21 days for a cycle(clinical use); 2) 125mg/m2 d1, 8, 15, 30 minutes intravenous injection, 28 days for a cycle(guideline recommand). Treatment to disease progression. The efficacy (CR, PR, SD, PD) is evaluated every 2-4 cycles.If the patient withdraws from the trial because he cannot tolerate the toxicity caused by one of the drugs, such as neurotoxicity or bone marrow toxicity, it is recommended to switch to other drugs and follow up to PFS and OS.Each group was planned to include 30 patients.

ELIGIBILITY:
Inclusion criteria

* Female, aged≥ 18 years old;
* Histopathologically confirmed HER-2 negative (definition: immunohistochemical IHC 0, or 1+, or in situ hybridization ISH, defined as the ratio of HER2 gene copy number to CEP17 signal number less than 2.0, or for single probe detection, HER2 gene copy number less than 6) in patients with recurrent or metastatic breast cancer;
* Up to two previous lines of chemotherapy were permitted for recurrent and metastatic diseases. And for endocrine therapy, the number of treatment lines can be omitted;
* With measurable lesions;
* The physical condition score of the Eastern American Cancer Collaboration Group (ECOG) was less than 1;
* Expected survival period>3 months;

Exclusion Criteria

* New York Heart Association NYHA scores identify patients with congestive heart failure at grade II or above;Uncontrolled brain metastasis;
* Patients with severe systemic infection;Patients with peripheral nerve injury of degree II or above, or known drug allergy or intolerance within 4 weeks before admission;
* Important organ disorders or diseases: liver and kidney dysfunction, history of myocardial infarction, unstable heart disease, chronic active hepatitis,etc;There is a history of other malignant tumors within 5 years (except cured cervical cancer or skin basal cell carcinoma);
* Patients who had received other antineoplastic treatments or other experimental drugs within one month before treatment;
* Patients who also participated in other clinical trials;
* Researchers believe that patients are not suitable for any medical condition to enter the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2019-02-21 (Actual); Primary Completion 2023-01-26 (Estimated); Study Completion 2023-01-26 (Estimated)

PRIMARY OUTCOMES:
PFS of two regimen | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  progession free survival and objective remission rate was put in to assessment after 2-4 cycle of treatment of either two regimen

SECONDARY OUTCOMES:
Side effect of two regimen | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  toxicity and tolerability would be evaluated after every cycle of treatment and will report a SAE within 24h

CONTACTS AND LOCATIONS:
Locations (1):
- BeijingCancerH, Haidian, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu Y, Song G, Di L, Jiang H, Ran R, Zhang R, Zhang Y, Li H. Three-Week Versus 4-Week Schedule of nab-Paclitaxel in Patients With Metastatic Breast Cancer: A Randomized Phase II Study. Oncologist. 2023 Dec 11;28(12):1102-e1302. doi: 10.1093/oncolo/oyad288. PMID 37882706